CLINICAL TRIAL: NCT01750476
Title: Modulation of Mucosal and Systemic Immunity by Hormonal Contraceptives
Status: Terminated | Type: Observational
Why Stopped: PI and lab have re-located study to The Ohio State University
Sponsor: Thomas Cherpes, DVM, MD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Thomas Cherpes, DVM, MD, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: PRO12010187; R01HD072663 (NIH)
Record Dates: First submitted 2012-12-10; First posted 2012-12-17 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Initiation of Oral Contraception (OC); Initiation of Depo-Provera (DMPA); Initiation of Mirena (LNG-IUD)
Keywords: oral contraception; Depo-Provera; Mirena
MeSH Terms: interventions — Levonorgestrel; Contraceptives, Oral; Medroxyprogesterone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Depo-Provera: Women who choose to initiate Depo-Provera
  Interventions: Drug: Depo-Provera
- Mirena: Women who choose to initiate Mirena (intrauterine device)
  Interventions: Drug: Mirena
- Oral contraception: Women who choose to initiate oral contraception
  Interventions: Drug: Oral contraception

INTERVENTIONS:
Drug: Mirena
  Groups: Mirena
Drug: Oral contraception
  Groups: Oral contraception
Drug: Depo-Provera
  Groups: Depo-Provera

SUMMARY:
The investigators are conducting a research study to understand how cells responsible for fighting infection (immune cells) are affected by hormonal contraceptive use. The investigators hypothesize that progestin-containing hormonal contraceptives (i.e., Depo-Provera) inhibit host response to infection. To test this hypothesis, the investigators will collect blood and genital tract samples from women before and after their initiation of a hormonal contraceptive (either birth control pills, Depo-Provera, or Mirena).

ELIGIBILITY:
Inclusion Criteria:

1. 15-25 years of age (inclusive)
2. History of regular menstrual cycle
3. Not pregnant
4. No plan to become pregnant in the next 3 months
5. Interested in beginning use of OC, DMPA, or LNG-IUD
6. Able to read and provide written informed consent (and consent from a parent/guardian if the participant is a minor)

Exclusion Criteria:

1. Anticipated move out of area that prevents return for a follow-up visit
2. Unavailability for follow-up visit
3. Less than 90 days post-partum or post-abortion
4. Sexually transmitted infection (STI) diagnosed less than 30 days prior to enrollment
5. Use of OC, contraceptive ring or patch, single rod implant, LNG-IUD, or copper-containing IUD less than 3 months prior to enrollment
6. DMPA injection less than 6 months prior to enrollment
7. History of immunosuppressive condition of current use of immunosuppressive medications
8. History of a cervical malignancy
9. Detection of cervical anatomic pathologic conditions that preclude cervical biopsy procurement
10. Intolerance or contradiction to use of OC, DMPA, or LNG-IUD

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women interested in initiating hormonal contraceptive use
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Proliferative capacity (i.e., ability to respond to antigen stimulation) of T cells isolated from the cervix of women before and after initiating a hormonal contraceptive | Prior to and ~ 1 month (but up to 2 months) after initiation of a hormonal contraceptive

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Cherpes, MD, Principal Investigator — assistant professor
Locations (1):
- UPMC Adolescent Clinic of Oakland, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Vicetti Miguel RD, Hendricks RL, Aguirre AJ, Melan MA, Harvey SA, Terry-Allison T, St Leger AJ, Thomson AW, Cherpes TL. Dendritic cell activation and memory cell development are impaired among mice administered medroxyprogesterone acetate prior to mucosal herpes simplex virus type 1 infection. J Immunol. 2012 Oct 1;189(7):3449-61. doi: 10.4049/jimmunol.1103054. Epub 2012 Aug 31. PMID 22942424
- [Background] Vicetti Miguel RD, Maryak SA, Cherpes TL. Brefeldin A, but not monensin, enables flow cytometric detection of interleukin-4 within peripheral T cells responding to ex vivo stimulation with Chlamydia trachomatis. J Immunol Methods. 2012 Oct 31;384(1-2):191-5. doi: 10.1016/j.jim.2012.07.018. Epub 2012 Jul 29. PMID 22850275